CLINICAL TRIAL: NCT03630757
Title: Effects of Manual Therapy on Pain, Spinal Mobility, Quality of Sleep and Emotional Status in Fibromyalgia Syndrome
Brief Title: Effects of Manual Therapy in Fibromyalgia Syndrome
Acronym: Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, TOMRIS DUYMAZ, Asst. Prof. Ph.D., Istanbul Bilgi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-40016-69
Record Dates: First submitted 2018-08-07; First posted 2018-08-15 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Fibromyalgia; Manual Therapies
Keywords: Fibromyalgia syndrome; Manual Therapies; Pain
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Patients were randomly divided into 2 groups of 20 people. A randomized list is prepared in a computer environment by a statistician for randomization. In this list, the odd numbers for the control group and the MT group were given double numbers. The group identification is printed on sequentially numbered cards placed in sealed envelopes. After enrollment, the numbered envelope was opened by the patient and the blind investigator. For the study group, manual therapy (MT) was given and the home exercise program was given and for the control group only home exercise program was given. In the study group, a total of 15 sessions of a manual therapy program including myofascial release and mobilization techniques were applied for 60-minute session for 3 weeks(5/wk). The treatment program has been implemented by a physiotherapist who specializes in this area.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): While holding the patient's head with the therapist's hands,the cervical spinous processes with the fingertips palpitate to the occipital condyle towards the proximal.Then the fingers of both hands applied pressure to the axis in the space between the occipital condyle and the spinous process
  Interventions: Other: Treatment
- Group 2 (Placebo Comparator): reaching to the feet while sitting together with warming and cooling periods
  Interventions: Other: Treatment

INTERVENTIONS:
Other: Treatment — In the study group, a total of 15 sessions of a manual therapy program including myofascial release and mobilization techniques were applied for 60-minute session for 3 weeks(5/wk).

SUMMARY:
Fibromyalgia syndrome (FMS) is among the most difficult diseases that restrict physical functions of patients due to persistent aches,sleep problems,psychological problems and decrease the quality of life. The aim of this study was to investigate the efficacy of manual therapy (MT) in the treatment of FMS patients.

DETAILED DESCRIPTION:
Fibromyalgia syndrome (FMS) etiology is a chronic musculoskeletal system characterized by widespread pain and hyperalgesia in the body that is not yet known. At the same time, FMS patients are accompanied by functional emotional disorders including persistent muscle soreness, muscle spasms, mood disorders such as chronic fatigue, sleep disturbances, paresthesia, morning stiffness, depression, and cognitive disorders. The prevalence in the general population in the world between 2-4%, but reaching up to 7% between 50-80 years of age the prevalence of a study conducted in Turkey were found to be 3.6%. Frequently seen in women between the ages of 40-60, the quality of life of patients with FMS falls because of generalized pain in their bodies, accompanied by stress in 30-45% of patients.

According to Chaitow, there are 3 factors in the etiology of the dysfunctional model of FMS syndrome (biochemical, biomechanical, psychosocial) : (1) Negative emotional state may cause specific biochemical change, weakening of immune functions and change in muscle tone (2) Hyperventilation, blood oxygenation at the neural level, general anxiety and anxiety state, change in the structural components of the thoracic and cervical region (3) Chemical changes in blood flow may cause emotional and structural changes. The neuroendocrine hypothalamic pituitary that controls primer stress response may have abnormal release of corticotropin releasing hormone, adrenocorticotropic hormone, and cortisol, which are part of the adrenal axis. Hypothalamic corticotropin releasing hormone delays corticotropin release by insufficiency of interleukin-6 regulation in the neuronal function defect. Although the pathophysiology is not yet fully understood, it is thought to be related to environmental and genetic factors. The basal autonomic status of FMS patients is characterized by increased sympathetic system and reduced parasympathetic system. The most basic complaints of patients are generalized pain. For this reason, peripheral and central nociceptive pathways are dominant in the view of being active in FMS patients. Intramuscular connective tissue dysfunction, myofascial tissue inflammation and fibroblasts and release of pro-inflammatory cytokines cause chronic peripheral sensitization in these patients. Some authors have reported that trigger points have central sensitization-inducing effects, while others have indicated that such a situation is not the case because the patient with each trigger point is not FMS. In recent biopsy studies, it has been found that the level of collagen in the endomyositis of the FMS muscles is increased, the production of N-carboxymethylsine, which is the oxidative stress marker, is increased, and the tissue damage is increased and the CD-68 positive macrophage levels in the interstitial tissue are increased in the muscles. The disturbance in the peripheral and central mechanisms leads to impairment of the postural control and therefore the increase in the frequency of falls with equilibrium losses. In the treatment of these symptoms, it was reported that the application of myofascial relaxation techniques had positive effects on patients' quality of life, sleep patterns, joint stiffness, neck and back pain.

Myofascial release therapy Myofascial relaxation restores pain relief by restoring soft-touch dysfunctions. Behind the therapeutic effects of myofascial relaxation is the effect on the connective tissue, that is, the fascia, one of the structures that play a fundamental role in the musculoskeletal functions. According to this theory, the facial system makes a great contribution to the different functions spreading from head to foot and to the dynamic movements of the body through its ability to move. Hardened and shortened facial tissue (due to recurrent micro trauma or acute injury), loss of functional capacity and pain due to reduced ability to shear. Myofascial relaxation therapy can also restore the mobility and pain sensation in the joints by stretching, loosening to the myofascial tissue. Myofascial relaxation therapy is a combination of manual traction and long stretching maneuvers to open facial adhesions. There are two basic myofascial release techniques, direct and indirect. In the direct relaxation technique, the therapist uses a hand or device to apply slight pressures (for 90-120 seconds) directly on the restricted tissue. The direct technique also includes self myofascial relaxation techniques. In the indirect technique, the myofascial complex is extended for a longer time under less load. With myofascial relaxation, normalization of the morphological and inflammatory responses of fibroblasts injured in the context of recurrent strains is possible.

The aim of this study was to investigate the efficacy of myofascial relaxation and mobilization techniques in the treatment of FMS patients on pain, trigger point number, FMS effect score, spinal mobility, sleep quality, anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 30 and 50
* No remission during the last 48 months
* Do not have regular physical activity
* Have had a daily activity limit of at least 1 day within 30 days

Exclusion Criteria:

* Cardiac, renal, hepatic insufficiency
* Severe physical disability
* Comorbid conditions (interstitial cystitis, inflammatory diseases)
* Chronic viral infection
* Fever
* Rheumatoid arthritis, herpes lupus
* Multiple sclerosis, polio, epilepsy
* Hypertension and hypotension
* Respiratory deficiencies during treatment
* Skin lesions
* Psychiatric disorders
* Past surgical history

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2018-07-07 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Baseline, up to 3 weeks
  The VAS pain score was measured to determine the pain level of the patients. The 0-10 cm chart was presented to the patient, with 0 no pain, 0 the most severe pain felt in life 10, 18 and was asked to mark the pain severity. Then the point marked with the millimetric ruler was measured and recorded.

SECONDARY OUTCOMES:
Pittsburgh Quality of Sleep Questionnaire Index | Baseline, up to 3 weeks
  This scale assesses sleep quality in the last month, the presence of sleep disturbance and the extent of this disorder. A total of 24 questions are covered, 19 of which are filled by the individual himself and 5 are filled by the individual's roommate. It is used only to evaluate the answers of the questions answered by the individual himself. Each item of the index takes a score between 0 (no annoyance) - 3 (serious annoyance). The sum of the scores of the seven subcomponents gives the total sleep quality score. The total score of the index is between 0 and 21, with scores below 5 indicating 'good' sleep quality and scores above 5 or 5 indicating 'poor' sleep quality.
Hospital of Anxiety and Depression Scale | Baseline, up to 3 weeks
  Developed by Zigmond and Snaith in 1983, scale is used to assess patients in terms of anxiety and depression. The HAD scale contains a total of 14 questions, seven of which measure anxiety and the other seven (double count) of depression. As a result of the validity and reliability studies performed by Aydemir et al., The cut-off score for the HAD anxiety score (HAD-A) was 10/11 and for the HAD depression score (HAD-D) it was 7/8. Accordingly, areas above these scores are considered at risk. The risk of anxiety and depression in HAD is self-assessment scale used to measure the level and change of violence.
Fibromyalgia Impact Questionnaire | Baseline, up to 3 weeks
  FIQ was used to assess functional status in a group of patients with fibromyalgia syndrome. This scale measures 10 different features including physical function, feeling good, not going to work, difficulty at work, pain, fatigue, morning fatigue, stiffness, anxiety and depression. Except for the ability to feel good, low scores indicate healing or less affected than 19 diseases. The FIQ is filled by the patient and takes about 5 minutes to complete. The maximum possible score for each descendant is 10. So the total maximum score is 100. While an average FMS patient has 50 points, more severely affected FMS patients usually score over 70 and 70 points.

CONTACTS AND LOCATIONS:
Overall Officials: TOMRIS DUYMAZ, Study Director — Istanbul Bilgi University
Locations (1):
- Istanbul Bilgi University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided